CLINICAL TRIAL: NCT00374166
Title: An Eight-week, Multicenter, Double-blind, Placebo- and Paroxetine-controlled Study Evaluating the Efficacy and Tolerability of Two Fixed Doses of SSR149415 (250 mg Bid and 100 mg Bid) in Outpatients With Generalized Anxiety Disorder
Brief Title: An Eight-week Study Evaluating the Efficacy and Tolerability of Two Doses of SSR149415 in Outpatients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI5880
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety Disorders
Keywords: Anti-anxiety agents; antidepressive agents; controlled clinical trial
MeSH Terms: conditions — Anxiety Disorders | interventions — 1-(5-chloro-1-((2,4-dimethoxyphenyl)sulfonyl)-3-(2-methoxyphenyl)-2-oxo-2,3-dihydro-1H-indol-3-yl)-4-hydroxy-N,N-dimethyl-2-pyrrolidinecarboxamide; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SSR149415 - 250 mg (Experimental): SSR149415 250 mg, twice daily for a maximum of 8 weeks
  Interventions: Drug: SSR149415
- SSR149415 - 100 mg (Experimental): SSR149415 100 mg and additional placebo capsules in order that all patients are being administered three capsules twice daily for a maximum of 8 weeks
  Interventions: Drug: SSR149415; Drug: Placebo
- Paroxetine (Active Comparator): Paroxetine 20 mg and additional placebo capsules in order that all patients are being administered three capsules twice daily for a maximum of 8 weeks
  Interventions: Drug: Placebo; Drug: Paroxetine
- Placebo (Placebo Comparator): Placebo for a maximum of 9 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSR149415 — Oral administration (capsules of 50 and 100 mg)
  Arms: SSR149415 - 100 mg; SSR149415 - 250 mg
Drug: Placebo — Oral administration (capsules)
  Arms: Paroxetine; Placebo; SSR149415 - 100 mg
Drug: Paroxetine — Oral administration (capsules)
  Arms: Paroxetine

SUMMARY:
The objective is to evaluate the efficacy and safety of two doses of SSR149415 (250 mg and 100 mg twice daily) compared to placebo and paroxetine 20 mg once daily in outpatients with generalized anxiety disorder

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized anxiety disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI) General Anxiety Disorder (GAD) Plus Module.

Exclusion Criteria:

* Total score of less than 22 on the (Hamilton Anxiety rating scale)HAM-A.
* Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than 17.
* Patients with a current history (within 6 months) of major depressive disorder or history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, antidepressants including Monoamine oxidase inhibitors (MAOIs) within 1 month, anxiolytics within 2 weeks, mood-stabilizer (lithium, anticonvulsants) within 1 month, and/or high dose or prolonged benzodiazepine (continuous use for 3 months prior to admission) use.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 56 in the 14-item Hamilton Anxiety Rating Scale (HAM-A) total score. | 8 weeks

SECONDARY OUTCOMES:
Change from baseline to Day 56 in the Clinical Global Impression (CGI) Severity of Illness score. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Griebel G, Beeske S, Stahl SM. The vasopressin V(1b) receptor antagonist SSR149415 in the treatment of major depressive and generalized anxiety disorders: results from 4 randomized, double-blind, placebo-controlled studies. J Clin Psychiatry. 2012 Nov;73(11):1403-11. doi: 10.4088/JCP.12m07804. Epub 2012 Oct 16. PMID 23146246